CLINICAL TRIAL: NCT07164742
Title: Pulmonary Rehabilitation to Reduce Post-Tuberculosis Morbidity (TB PURE) A Randomized Multi-Centre Trial
Brief Title: Parent Study Name: Pulmonary Rehabilitation to Reduce Post-Tuberculosis Morbidity (TB Pure)
Acronym: TB Pure
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB00412142; 1R01AI169588-01A1 (NIH)
Record Dates: First submitted 2025-09-02; First posted 2025-09-10 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: TB - Tuberculosis; TB; TB Infection
Keywords: pulmonary tuberculosis; Pulmonary Rehabilitation; post-tuberculosis respiratory morbidity; Drug-sensitive TB
MeSH Terms: conditions — Latent Tuberculosis; Tuberculosis, Pulmonary

STUDY DESIGN:
Intervention Model Description: Individual-level, unblinded randomized controlled trial of an 8-week (short arm) or 24-week (extended arm) pulmonary rehabilitation program, relative to standard of care, to prevent post-tuberculosis respiratory morbidity. Randomization will occur in a 1:1:1 ratio at the initiation of treatment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Short Arm Intervention (Experimental): 8 weeks (short arm) of a pulmonary rehabilitation (PR) program
  Interventions: Behavioral: 8 week (short arm) Intervention - pulmonary rehabilitation
- Long Arm Intervention (Experimental): 24 weeks (extended arm) of a pulmonary rehabilitation (PR) program
  Interventions: Behavioral: 24 week (long arm) Intervention - pulmonary rehabilitation
- Standard of care (No Intervention): Standard TB treatment without specific pulmonary rehabilitation

INTERVENTIONS:
Behavioral: 8 week (short arm) Intervention - pulmonary rehabilitation — 8 weeks (short arm) of a pulmonary rehabilitation (PR) program, administered during TB treatment, comprising of exercise training, counselling and education, and airway clearance techniques.
  Arms: Short Arm Intervention
Behavioral: 24 week (long arm) Intervention - pulmonary rehabilitation — 24 weeks (extended arm) of a pulmonary rehabilitation (PR) program, administered during TB treatment, comprising of exercise training, counselling and education, and airway clearance techniques.
  Arms: Long Arm Intervention

SUMMARY:
Individual-level, unblinded randomized controlled trial of an 8-week (short arm) or 24-week (extended arm) pulmonary rehabilitation program, relative to standard of care, to prevent post-tuberculosis respiratory morbidity. Randomization will occur in a 1:1:1 ratio at the initiation of treatment.

DETAILED DESCRIPTION:
8 weeks (short arm) or 24 weeks (extended arm) of a pulmonary rehabilitation (PR) program, administered during TB treatment, comprising of exercise training, counselling and education, and airway clearance techniques.

Objectives:

1. To compare the effectiveness of two home-based PR programs, administered during TB treatment, for preventing post-TB respiratory morbidity.
2. To describe the intersection between clinic-level service organization, fidelity of intervention delivery, and change in client behavior for the two PR programs.
3. To compare the costs, cost-effectiveness, and budget impact of the two different PR strategies implemented as a routine program.

ELIGIBILITY:
Inclusion Criteria:

* Age at least 18 years
* Microbiologically confirmed (smear microscopy, GeneXpert or culture) pulmonary TB disease*
* Not completed more than 2 weeks of TB treatment
* Receiving TB care at the outpatient clinics at the TB PuRe study sites
* Willingness to complete 48 weeks of study evaluations.
* Access to a smartphone.

Exclusion Criteria:

* Modified Medical Research Council score of 0 points (dyspnea only with strenuous exercise)
* Multi or extensively drug-resistant TB disease*
* Extrapulmonary TB disease at any clinical sites without pulmonary involvement
* TB meningitis or TB of the spine
* Symptomatic cardiovascular disease, including coronary artery disease, arrhythmias and congestive cardiac failure.
* Karnofsky Score < 40 points
* Any medical condition that prevents pulmonary rehabilitation eg: fracture of lower/upper limbs/pregnancy
* Bronchodilators and/or corticosteroids inhaled or otherwise.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 690 (Estimated)
Dates: Start 2026-02-15 (Estimated); Primary Completion 2028-09-15 (Estimated); Study Completion 2028-09-15 (Estimated)

PRIMARY OUTCOMES:
Six-Minute Walk Test (6MWT) distance (meters) | 48 weeks post enrollment
  Mean distance compared between study arms

SECONDARY OUTCOMES:
Six minute walk test (6MWT) distance (meters) | 8,16 & 24 weeks post enrollment
  Mean 6MWT distance compared between study arms at 8,16 & 24 weeks after enrollment.
Absolute percent change in Mean Six minute walk test (6MWT) distance | 8,16, 24 & 48 weeks post enrollment
  Difference between study arms in the absolute and percent change in mean 6MWT distance
Proportion of Participants with change in Six minute walk test (6MWT) distance (meters) | 8,16, 24 & 48 weeks post enrollment
  Difference between study arms in the proportion of participants with an Minimal Clinically Important Difference (MCID) change in the 6MWT distance
St. George's Respiratory Questionnaire (SGRQ) score | 8,16,24 & 48 weeks post enrollment
  The questionnaire measures respiratory health quality of life in three areas with a total score ranging from 0-100. A higher score indicates poorer health status.
Absolute change in score for St. George's Respiratory Questionnaire (SGRQ) | 8,16,24 & 48 weeks post enrollment
  Difference between study arms in the absolute change in questionnaire score
Percent change in score for St. George's Respiratory Questionnaire (SGRQ) | 8,16,24 & 48 weeks post enrollment
  Difference between study arms in the percent change in questionnaire score
Proportion of participants with change in score for St. George's Respiratory Questionnaire (SGRQ) | 8,16,24 & 48 weeks post enrollment
  Difference between study arms in the proportion of participants with an MCID change in questionnaire score
Modified Medical Research Council (mMRC) Dyspnoea Scale | 8,16,24 & 48 weeks post enrollment
  The Modified Medical Research Council Dyspnea Scale scores range from 0 (minimum) to 4 (maximum), with higher scores indicating more severe dyspnea.
Absolute change in the Modified Medical Research Council (mMRC) Dyspnoea Scale | 8,16,24 & 48 weeks post enrollment
  Difference between study arms in the absolute change in questionnaire score
Percent change in the Modified Medical Research Council (mMRC) Dyspnoea Scale | 8,16,24 & 48 weeks post enrollment
  Difference between study arms in the percent change in questionnaire score
Proportion of participants with change in Modified Medical Research Council (mMRC) Dyspnoea Scale | 8,16,24 & 48 weeks post enrollment
  Difference between study arms in the proportion of participants with an MCID change in questionnaire score
Chronic Respiratory Disease Questionnaire (CRQ) Dyspnea score | 8,16,24 & 48 weeks post enrollment
  The CRQ assesses dyspnea on a Likert scale from 1 (Extremely short of breath) to 7 (Not at all short of breath). Total score ranges from 5 - 35. Lower scores indicate higher severity of dyspnea.
Absolute change in Chronic Respiratory Disease Questionnaire (CRQ) Dyspnea score | 8,16,24 & 48 weeks post enrollment
  Difference between study arms in the absolute change in questionnaire score
Percent Change in Chronic Respiratory Disease Questionnaire (CRQ) Dyspnea score | 8,16,24 & 48 weeks post enrollment
  Difference between study arms in the percent change in questionnaire score
Proportion of participants with change in Chronic Respiratory Disease Questionnaire (CRQ) Dyspnea sore | 8,16,24 & 48 weeks post enrollment
  Difference between study arms in the proportion of participants with an MCID change in questionnaire score
COPD Assessment Test (CAT) score | 8,16,24 & 48 weeks post enrollment
  CAT total score range is from 0-40, higher scores indicates a more severe impact of COPD on a patient's life.
Absolute change in COPD Assessment Test (CAT) score | 8,16,24 & 48 weeks post enrollment
  Difference between study arms in the absolute change in questionnaire score
Percent change in COPD Assessment Test (CAT) score | 8,16,24 & 48 weeks post enrollment
  Difference between study arms in the percent change in questionnaire scores 8,16, 24 & 48 weeks after enrollment.
Proportion of participants with a change in COPD Assessment Test (CAT) score | 8,16,24 & 48 weeks post enrollment
  Difference between study arms in the proportion of participants with an MCID change in questionnaire score
FEV1 volume (mL) - Lung function | 24 & 48 weeks post enrollment
  FEV1 volume (mL) compared between study arms at 24 & 48 weeks after enrollment.
Absolute change in FEV1 volume (mL) - Lung function | 8, 16, 24 & 48 weeks post enrollment
  Difference between study arms in the absolute change in FEV1 volume
Percent change in FEV1 volume (mL) - Lung function | 8, 16, 24 & 48 weeks post enrollment
  Difference between study arms in the percent change in FEV1 volume by 8,16, 24 & 48 weeks after enrollment.
Proportion of participants with change in FEV1 and/or FVC volume (mL) - Lung function | 8, 16, 24 & 48 weeks post enrollment
  Difference between study arms in the proportion of participants with a MCID change in FEV1 and/or FVC
FVC volume (mL) - Lung function | 24 & 48 weeks post enrollment
  FVC volume (mL) compared between study arms
Absolute change in FVC volume (mL) - Lung function (FEV1 and FVC) | 8,16, 24 & 48 weeks post enrollment
  Difference between study arms in the absolute change in FVC volume
Percent change in FVC volume (mL) - Lung function (FEV1 and FVC) | 8,16, 24 & 48 weeks post enrollment
  Difference between study arms in the percent change in FVC volumes

OTHER OUTCOMES:
Proportion of participants experiencing unfavorable treatment outcomes (Exploratory Outcome Measure) | 4, 8,12, 16, 20, 24, & 48 weeks post enrollment
  Arm comparisons of the proportion of participants experiencing any unfavorable TB treatment outcome of failure, recurrence, or death

CONTACTS AND LOCATIONS:
Overall Officials: Akshay Gupte, PhD MBBS MSPH, Principal Investigator — Boston University; Jonathan Golub, PhD MPH, Principal Investigator — Johns Hopkins University

IPD SHARING:
Plan to Share IPD: No